CLINICAL TRIAL: NCT06803212
Title: Effect of Dual-Task Interference on Upper Extremity Motor Experience With Parkinson's Disease
Brief Title: Investigation of Dual-Task Exercise's Effect in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emre Şenocak (Other)
Responsible Party: Sponsor-Investigator, Emre Şenocak, Assistant Professor (PhD), Karadeniz Technical University
Organization: Karadeniz Technical University (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2024/109
Record Dates: First submitted 2025-01-27; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Therapy (Active Comparator): This group were performed just conventional physiotherapy.
  Interventions: Other: Conventional Physiotherapy Program
- Dual-Task Interference (Experimental): Dual-task exercises were applied during conventional physiotherapy practices.
  Interventions: Other: Conventional Physiotherapy Program; Other: Dual-Task Interference

INTERVENTIONS:
Other: Conventional Physiotherapy Program — The patients' conventional physiotherapy program included stretching, strengthening, balance, and coordination exercises according to their individual needs
Other: Dual-Task Interference — This intervention consisted of counting backward, reading words backward, and remembering word exercises.
  Arms: Dual-Task Interference

SUMMARY:
This study was conducted to investigate the effects of dual-task training on upper extremity motor functions in patients with Parkinson's disease. A total of 32 patients participated in the study. Patients were divided into two groups by randomization. One group received only conventional physiotherapy applications, while the other group performed dual-task exercises in addition. Dual-task exercises were performed while conventional treatment was applied. The treatment program was applied as 60x5x6 min/day/week.

Conventional treatment was determined according to the individual needs of the patients, including the lower and upper extremities. Dual-task interventions included performing such as counting backward, word recall, and reading words backward.

Assessments were repeated twice: Baseline and after a 30-session. "Demographic Information", "Movement Disorder Society (MDS)-Unified Parkinson's Disease Rating Scale (MDS-UPDRS)", "Box and Block Test" and "Parkinson Disease Questionnaire (PDQ-39) were used as assessment tools.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 50-85 years with a diagnosis of Stage 1-3 Parkinson's disease, based on the Hoehn & Yahr Scale
* Patients had to have no issues with performing basic mathematical operations, - A Mini-Mental State Examination (MMSE) score above 24 points,
* Regular medication use for at least 4 weeks (for patients who were prescribed medical treatment),
* No comorbid neurological, neuromuscular, or orthopedic diseases

Exclusion Criteria:

* Patients with vision or hearing impairments,
* Moderate-to-severe fluctuations in tremor or dyskinesia,
* Having deep brain stimulator implants, or sensory loss in the upper extremities.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2024-06-28 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Movement Disorder Society (MDS)-Unified Parkinson's Disease Rating Scale (MDS-UPDRS): | Baseline of the study
  The scale consists of four separate domains. The first section includes non-motor experiences in daily life (13 items), the second section includes motor experiences in daily life (13 items), the third section involves motor examination (33 items), and the last section addresses motor complications (6 items). The scale contains 65 individual items in total. Items are generally scored between 0-4, with some Yes/No items. The domains of the scale directly related to the upper extremities, including eating, dressing, cleaning, writing, rigidity, finger movements, hand movements, pronation and supination of the hand, postural tremor in the hands, kinetic tremor in the hands, resting tremor, and tremor persistence, were used in this study (Figure 1). The MDS-UPDRS scoring was performed while patients were in the "ON" state.
Movement Disorder Society (MDS)-Unified Parkinson's Disease Rating Scale (MDS-UPDRS): | End of the 30th physiotherapy session
  The scale consists of four separate domains. The first section includes non-motor experiences in daily life (13 items), the second section includes motor experiences in daily life (13 items), the third section involves motor examination (33 items), and the last section addresses motor complications (6 items). The scale contains 65 individual items in total. Items are generally scored between 0-4, with some Yes/No items. The domains of the scale directly related to the upper extremities, including eating, dressing, cleaning, writing, rigidity, finger movements, hand movements, pronation and supination of the hand, postural tremor in the hands, kinetic tremor in the hands, resting tremor, and tremor persistence, were used in this study (Figure 1). The MDS-UPDRS scoring was performed while patients were in the "ON" state.

SECONDARY OUTCOMES:
Box Block Test (BBT) | Baseline of the study
  The BBT consists of a panel and two boxes, one containing 150 wooden blocks. The patient is asked to transfer blocks from one box to another within 60 seconds, one block at a time, using only one hand. The test is repeated with both hands. The number of blocks moved provides the total score. A higher score indicates better manual dexterity.
Box Block Test (BBT) | End of the 30th physiotherapy session
  The BBT consists of a panel and two boxes, one containing 150 wooden blocks. The patient is asked to transfer blocks from one box to another within 60 seconds, one block at a time, using only one hand. The test is repeated with both hands. The number of blocks moved provides the total score. A higher score indicates better manual dexterity.
Parkinson's Disease Questionnaire - 39 (PDQ-39) | Baseline of the study
  This licensed tool assesses the quality of life associated with Parkinson's disease with a total of 39 items. Each item is scored between 0-4, with higher scores indicating poor quality of life. Responses are converted into hundredths for scoring, and the total score ranges from 0 to 100 points.
Parkinson's Disease Questionnaire - 39 (PDQ-39) | End of the 30th physiotherapy session
  This licensed tool assesses the quality of life associated with Parkinson's disease with a total of 39 items. Each item is scored between 0-4, with higher scores indicating poor quality of life. Responses are converted into hundredths for scoring, and the total score ranges from 0 to 100 points.
Demographic Data Form | Baseline of the study
  This form was developed by the investigators and included age, body mass index, disease duration, sex, dominant limb, education level, presence of freezing, presence of tremor, MMSE score, total daily dose of levodopa, and Hoehn & Yahr Staging.

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul Tıp Merkezi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No